CLINICAL TRIAL: NCT05352555
Title: Comparison of Treatment Efficacy of Automated Robotic Maneuvering System (RMS) Reposition Chair Versus Traditional Manual Repositioning Maneuvers in Benign Paroxysmal Positional Vertigo (BPPV)
Brief Title: Automated Robotic Maneuvering System (RMS) vs Manual Reposition Maneuver in Treatment of Benign Paroxysmal Positional Vertigo (BPPV)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stratejik Yenilikci Girisimler Ltd. (Industry)
Collaborators: Haseki Sultangazi Teaching and Research Hospital, University of Health Sciences (Unknown)
Responsible Party: Principal Investigator, Murat Haluk Ozkul, Chief Medical Officer (CMO), Stratejik Yenilikci Girisimler Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYG-RMS-18
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Automated; Robotic; Vertigo; Epley maneuver; RMS chair; Reposition chair; Dizziness; Vestibular diseases; Multi canal BPPV
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Patients previously diagnosed with BPPV were referred to vestibular laboratory at the Department of Otolaryngology at Haseki Sultangazi Teaching and Research Hospital. Videonystagmography was performed on all subjects to confirm the BPPV diagnosis. Patients were then randomly divided into two groups; experimental and control. The experimental group was treated with RMS, while control group was treated with traditional manual canalith repositioning maneuvers on an examination table.
Who Masked: Participant, Care Provider
Masking Description: Every enrolled patients records were randomized, and based on the outcome, subjects were either assigned to control or experimental arm groups. A report detailing the outcome, but omitting the method of treatment, was given to patients and their care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Maneuvering System (RMS) (Experimental): BPPV subtype diagnosis and corresponding treatment will be performed using automated RMS chair and recorded with video frenzel goggle.
  In cases of posterior canal involvement, Epley's maneuver will be used for canalithiasis and cupulolithiasis. Semont maneuver will be used as a second-line treatment for cupulolithiasis, in cases of initial failure.
  In cases of horizontal canal involvement, Barbecue (Lempert) maneuver will be used. If canalithiasis or cupulolithiasis is diagnosed, Gufoni's maneuver will be performed.
  In cases of anterior canal involvement, Yacovino's maneuver will be used.
  Interventions: Device: Automated vertigo repositioning chair
- Canalith Reposition Maneuver (Active Comparator): BPPV subtype diagnosis and corresponding treatment will be performed with manual repositioning maneuvers and recorded with video frenzel goggle.
  In cases of posterior canal involvement, Epley's maneuver will be used. In cases of horizontal canal involvement, Log roll maneuver will be used. In cases of anterior canal involvement, Yacovino's maneuver will be used.
  Interventions: Other: Canalith Reposition Maneuver

INTERVENTIONS:
Device: Automated vertigo repositioning chair — Patients are strapped to the chair with a safety harness, and video fenzel goggle are worn.
  Automated diagnostic procedures are performed to determine vertigo subtype and orientation (Left/Right) (described below).
  1. Dix-Hallpike (for posterior canal involvement)
  2. Supine roll (for horizontal canal involvement)
  3. (Optional) Deep Head Hanging (for anterior canal involvement)
  If nystagmus is detected during automated diagnostic maneuvers, BPPV subtype is diagnosed, and corresponding automated treatment maneuver will be performed (described below).
  1. Epley's and/or Semont's maneuver (for posterior canal involvement)
  2. Barbecue and/or Gufoni's maneuver (for horizontal canal involvement)
  3. Yacovino's maneuver (for anterior canal involvement)
  10 minutes after performing automated treatment maneuver, provocative diagnostic test maneuver was performed once again to ensure successful intervention.
  A follow-up was done one week later at the earliest.
  Other Names: Robotic Maneuvering System (RMS)
  Arms: Robotic Maneuvering System (RMS)
Other: Canalith Reposition Maneuver — Patients were seated on a examination table and given videonystagmography goggles (VNG).
  Manual diagnostic procedures are performed to determine vertigo subtype and orientation.
  The manual diagnostic procedures for Left and Right sided semicircular canals are:
  1. Dix-Hallpike (for posterior canal involvement)
  2. Supine roll and Bow and Lean (for horizontal canal involvement)
  If nystagmus is detected during diagnostic maneuvers, BPPV subtype is diagnosed, and corresponding treatment maneuvers will be performed manually.
  The automated treatment maneuvers are:
  1. Epley's maneuver (for posterior canal involvement)
  2. Barbecue and/or Gufoni's maneuver (for horizontal canal involvement)
  Patients were called back for a follow up 2 days after performing manual treatment maneuvers. Provocative diagnostic testing maneuvers were performed again to ensure successful intervention.
  A second follow-up was done one week later at the earliest.
  Other Names: Manual Reposition Maneuver
  Arms: Canalith Reposition Maneuver

SUMMARY:
Comparison of treatment efficacy of an automated robotic maneuvering system (RMS) repositioning chair versus manual positioning maneuvers in Benign Paroxysmal Positional Vertigo.

DETAILED DESCRIPTION:
The standard treatments for Benign Paroxysmal Positional Vertigo (BPPV) are manual positioning maneuvers. This method, beyond being costly and requiring extensive training, is a significant burden on healthcare resources. We developed an automated robotic maneuvering system, hereby known as RMS, to tackle this problem. Our Clinical Investigation is two-fold; (1) test the safety of RMS and, (2) understand the viability of RMS for treating BPPV when compared to manual positioning maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Characteristic positional nystagmus (for BPPV)
* Positive Dix-Hallpike
* Positive supine roll test
* Positive Deep Head Hanging
* Vertigo-Dizziness Imbalance symptom scores compatible with BPPV

Exclusion Criteria:

* Pregnant patients
* Patients who have taken vertigo suppressing agents (Dimenhydrinate) in the last 48 hours
* Patients taller than 200 cm (2.0 m)
* Patients who have had a cardiovascular or neurosurgical operation in the last month
* Patients with retinal detachment and/or glaucoma
* Lack of treatment cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Treatments | 1 month (30 days)
  Number of treatment necessary to achieve resolution of vertigo and nystagmus
Treatment success | After treatment: 1 week - 1 month (30 days)
  Number of subjects achieving resolution of vertigo and nystagmus after one treatment

SECONDARY OUTCOMES:
Vertigo-Dizziness Imbalance (VDI) questionnaire | 1 month (30 days)
  Comparison of pre-treatment and post-treatment score based on symptoms and quality of life
Adverse events | 1 month (30 days)
  Registration of adverse events and safety issues related to RMS.

CONTACTS AND LOCATIONS:
Overall Officials: Murat H Ozkul, M.D., Principal Investigator — StatejikYG
Locations (1):
- Haseki Sultangazi Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan J, Yu D, Feng Y, Song Q, You J, Shi H, Yin S. Comparative study of the efficacy of the canalith repositioning procedure versus the vertigo treatment and rehabilitation chair. Acta Otolaryngol. 2014 Jul;134(7):704-8. doi: 10.3109/00016489.2014.899711. Epub 2014 May 7. PMID 24807849
- [Background] Choung YH, Shin YR, Kahng H, Park K, Choi SJ. 'Bow and lean test' to determine the affected ear of horizontal canal benign paroxysmal positional vertigo. Laryngoscope. 2006 Oct;116(10):1776-81. doi: 10.1097/01.mlg.0000231291.44818.be. PMID 17003735
- [Background] West N, Hansen S, Moller MN, Bloch SL, Klokker M. Repositioning chairs in benign paroxysmal positional vertigo: implications and clinical outcome. Eur Arch Otorhinolaryngol. 2016 Mar;273(3):573-80. doi: 10.1007/s00405-015-3583-z. Epub 2015 Mar 7. PMID 25749489
- [Background] Bhattacharyya N, Baugh RF, Orvidas L, Barrs D, Bronston LJ, Cass S, Chalian AA, Desmond AL, Earll JM, Fife TD, Fuller DC, Judge JO, Mann NR, Rosenfeld RM, Schuring LT, Steiner RW, Whitney SL, Haidari J; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: benign paroxysmal positional vertigo. Otolaryngol Head Neck Surg. 2008 Nov;139(5 Suppl 4):S47-81. doi: 10.1016/j.otohns.2008.08.022. PMID 18973840
- [Background] Pedersen MF, Eriksen HH, Kjaersgaard JB, Abrahamsen ER, Hougaard DD. Treatment of Benign Paroxysmal Positional Vertigo with the TRV Reposition Chair. J Int Adv Otol. 2020 Aug;16(2):176-182. doi: 10.5152/iao.2020.6320. PMID 32784154
- [Background] Nakayama M, Epley JM. BPPV and variants: improved treatment results with automated, nystagmus-based repositioning. Otolaryngol Head Neck Surg. 2005 Jul;133(1):107-12. doi: 10.1016/j.otohns.2005.03.027. PMID 16025062
- [Background] Richard-Vitton T, Seidermann L, Fraget P, Mouillet J, Astier P, Chays A. [Benign positional vertigo, an armchair for diagnosis and for treatment: description and significance]. Rev Laryngol Otol Rhinol (Bord). 2005;126(4):249-51. French. PMID 16496552
- [Background] Yanik B, Kulcu DG, Kurtais Y, Boynukalin S, Kurtarah H, Gokmen D. The reliability and validity of the Vertigo Symptom Scale and the Vertigo Dizziness Imbalance Questionnaires in a Turkish patient population with benign paroxysmal positional vertigo. J Vestib Res. 2008;18(2-3):159-70. PMID 19126986